CLINICAL TRIAL: NCT05917873
Title: Metabolic Effects of Four-week Lactate-ketone Ester Supplementation
Acronym: MetaLaKe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry); Aarhus University Hospital (Other); Riisfort (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 98128
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Insulin sensitivity; Lipolysis; Appetite
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LaKe arm (Experimental): Ingestion of a combined lactate and ketone body ester, 25 ml twice daily for 28 days.
  Interventions: Dietary Supplement: LaKe Ester
- Placebo arm (Placebo Comparator): Placebo treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LaKe Ester — Lactate and ketone body ester (one equivalent of S-lactate and one equivalent of 1,3-butanediol / D-β-hydroxybutyrate)
  Arms: LaKe arm
Dietary Supplement: Placebo — Taste and appearance matched noncaloric placebo
  Arms: Placebo arm

SUMMARY:
Recent research reveals intriguing results concerning the role of exogenous lactate and the ketone body 3-hydroxybutyrate (3-OHB) as therapeutic tools to combat obesity and related conditions. Thus, oral administration of lactate and 3-OHB have separately been shown to suppress appetite sensations and slow gastric emptying while administered orally. Both seem to inhibit lipolysis while oral 3-OHB administration have shown direct insulin sensitizing effects. Furthermore, both substrates can be used as fuel for the heart.

The goal of this placebo-controlled randomized crossover design is to test exogenous lactate and the ketone body 3-hydroxybutyrate (3-OHB) in healthy, non-diabetic, obese adults.

The main questions it aims to answer are if chronic administration of LaKe ester affect or improve the following endpoints:

* Insulin sensitivity
* Appetite sensations
* Gastric emptying
* Lipolysis
* Cardiac output
* Left Ventricular Ejection Fraction
* Global Longitudinal Strain and other echocardiographic measures listed below

Participants will ingest a combined lactate and ketone body ester (LaKe ester) or placebo twice a day for 28 days before experimental days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-60 years
* BMI range 30-40
* Glycated haemoglobin (HbA1c) < 48 mmol/mol
* Otherwise 'healthy'
* Written and oral consent

Exclusion Criteria:

* Medication that affect energy or glucose metabolism, eg metformin, insulin or Glucagon-like peptide-1 receptor (GLP-1) agonists
* Specific diets (eg practicing ketogenic diets)
* Cardiac arrhythmias (eg atrial fibrillation)
* Ongoing acute/chronic serious diseases (eg, anemia, chronic kidney or liver disease)
* Inability to understand Danish or English

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity expressed as an M-value | Throughout the cross-over design, approximately 12 weeks
  On all study days, a hyperinsulinemic-euglycemic clamp is used to determine insulin sensitivity: continuous infusion of insulin (1 milliunit · kg lean body mass-1 · min-1) for 2 hours. The blood glucose is clamped at 5 mmol/l.

SECONDARY OUTCOMES:
Differences in lipolysis rate | Throughout the cross-over design, approximately 12 weeks
  Measured as differences in palmitate flux
Differences in body weight and composition | Throughout the cross-over design, approximately 12 weeks
  Dual-energy X-ray absorptiometry (DEXA) scan to assess total fat mass (kg), lean body mass (kg), and bone mass (kg)
Differences in gastric emptying rate | Throughout the cross-over design, approximately 12 weeks
  Evaluated by using the acetaminophen test
Cardiac Output (CO) | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes in left ventricular outflow tract (LVOT), velocity time integral (VTI) and heart rate (HR)
Left Ventricular Ejection Fraction (LVEF) | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes
Tricuspid annular plane systolic excursion (TAPSE) | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes
Global Longitudinal Strain (GLS) | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes
Mitral inflow velocities (E and A) | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes
Mitral plane velocities in the lateral mitral annulus (e' and s') | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes
Global work index (GWI) | Throughout the cross-over design, approximately 12 weeks
  Echocardiographic changes
Changes in blood concentrations of 3-OHB | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of lactate | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of free fatty acids | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of glucose | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of insulin | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in plasma concentrations of growth/differentiation factor 15 (GDF-15) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of gastric inhibitory polypeptide (GIP) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of ghrelin | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of glucagon | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of liver-expressed antimicrobial peptide 2 (LEAP-2) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of C-peptide | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of triglycerides | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of cholesterol | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of brain-derived neurotrophic factor (BDNF) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of N-lactoyl-phenylalanine (Lac-Phe) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Fibrosis-4 (FIB-4) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling of alanine aminotransferase (ALAT), aspartate transaminase (ASAT), and thrombocytes
Changes in blood concentrations of erythrocyte volume fraction (EVF) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of Erythropoietin (EPO) | Throughout the cross-over design, approximately 12 weeks
  Blood sampling
Changes in blood concentrations of inflammation markers | Throughout the cross-over design, approximately 12 weeks
  Blood sampling of C reactive protein (CRP) and leucocytes
Mood, assessed by Major Depression Inventory score (MDI) | Throughout the cross-over design, approximately 12 weeks
  Change in MDI score measured by Major Depression Inventory. The theoretical sum score ranges from 0 (no depression) to 50 (maximum depression).
Anxiety Symptom Scale questionnaire (ASS) | Throughout the cross-over design, approximately 12 weeks
  Change in the Anxiety Symptom Scale questionnaire to screen for anxiety disorders. The theoretical sum score ranges from 0 (no anxiety) to 60 (maximum anxiety).
Supplement tolerability | Throughout the cross-over design, approximately 12 weeks
  Assessed using a symptom questionnaire covering every organ system, including GI symptoms measured through the validated "Beverage Tolerability Questionnaire". Participants will rate the frequency of each item on a scale from 0 (no symptoms) to 5 (severe symptoms).
Control of Eating Questionnaire (CoEQ) | Throughout the cross-over design, approximately 12 weeks
  The CoEQ has been used in clinical trials as a multi-dimensional measure of appetite, craving and mood regulation. Based on the previous 7 days, subjects will be asked to answer 21 questions (20 rated on a 100 mm visual analogue scale and one open-ended).

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Denmark

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT05917873/SAP_001.pdf